CLINICAL TRIAL: NCT03609086
Title: Investigation of Melatonin Production in Pregnancy: a Pilot Study to Define the Contribution of the Placenta
Brief Title: Melatonin in Pregnancy
Acronym: MEL-P2
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-020-18
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Melatonin analysis — Measurement of 6-hydroxymelatonin

SUMMARY:
Melatonin is well known for its role in the sleep-wake cycle and is synthesised in response to low light levels from the pineal gland. In our previous study it was found that serum melatonin levels increased dramatically during pregnancy, such that levels were up to 100 fold higher in the third trimester compared to healthy non-pregnant women. The placenta contains the enzymes which are involved in synthesising melatonin but it is unclear if this is the source of the high levels in pregnancy. Severe pre-eclampsia has been reported to be associated with low levels of melatonin. In this study its is proposed to measure serum melatonin immediately before and after delivery and in cord blood and relate the levels to those in the placenta itself. This will contribute to the potential role for melatonin as a biomarker for obstetric disease and potentially as a therapeutic agent in future. This observational pilot study aims to measure serum and placental melatonin levels (as the major metabolite 6-hydroxymelatonin sulphate) in pregnant women undergoing elective Caesarean section.

DETAILED DESCRIPTION:
Background Melatonin, a substance produced by the pineal gland, is well known for its role in the sleep-wake cycle but it is less well known as an effective antioxidant. It is able to access all parts of the cell, and can cross the blood-brain and placental barrier.

Melatonin has been reported to be synthesised in the placenta and may have both receptor mediated and non-receptor mediated protective functions during pregnancy. Severe pre-eclampsia has been reported to be associated with low levels of melatonin in the placenta although it is not known if the placental melatonin contributes to circulating levels.1,2 Despite this, melatonin levels have been proposed as a biomarker of pre-eclampsia. More information on the role of melatonin and metabolism of melatonin in pregnancy would inform planning of larger research studies to investigate the potential role for melatonin as a bio-marker for obstetric disease and potentially as a therapeutic agent in future.

Melatonin is synthesized endogenously from serotonin via two steps; the first, rate limiting step is arylalkylamine N-acetyltransferase mediated acetylation of serotonin to N-acetyl serotonin. The second step is methylation of N-acetyl serotonin via the enzyme hydroxyindole O-methyltransferase (also called N-acetylserotonin O-methyl-transferase).3,4 Interrogation of our database of next generation sequencing analysis of 80 human foetal livers revealed that the genes encoding these enzymes were not present although those encoding related acetyltransferases were. We can conclude that the human foetal liver is not a site of melatonin synthesis.

Our previous work found melatonin levels do however increase markedly during pregnancy and are up to 50-100 times higher than non-pregnant women in the third trimester (Figure). The physiological role of these elevated melatonin levels remains a supposition and the relationship of melatonin levels in the placenta with the maternal and foetal circulations at different stages of pregnancy are unclear. Melatonin synthesizing enzymes have been found in human placental tissue, however it is not clear whether placental production of melatonin is directly related to the elevated circulating maternal melatonin levels.

The production of melatonin is catalysed by specific enzymes and although these enzymes have been found in placental tissue, it is not known if the high melatonin levels in pregnancy come from the placenta and what the role of this melatonin is. It is proposed to measure melatonin in placentas and maternal/cord blood from women undergoing planned Caesarean section. The results should enable defining as to whether the placenta is a major source of melatonin and how the pattern of production changes in pregnancy. The blood samples taken from women having a Caesarean section and the umbilical cord will provide information about the role of melatonin at delivery.

If melatonin levels in the maternal circulation falls after delivery and placental tissue melatonin levels are well above limits of detection, then a firm conclusion that the placenta is the source of elevated maternal melatonin would be justified. This observational pilot study aims to measure 6-hydroxymelatonin sulphate levels in blood from women undergoing Caesarean section and umbilical cords, and from placental tissue.

This is an observational pilot study to investigate 6-hydroxymelatonin sulphate levels in blood from pregnant women immediately before and after delivery, from umbilical cord blood at the time of delivery and in samples of placental tissue.

Healthy pregnant women will be recruited at the pre-Caesarean section pre-assessment clinic.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective caesarian section
* Singleton pregnancy
* Aged 16-45
* Taking no regular medication other than pregnancy related vitamins or supplements

Exclusion Criteria:

* Pregnancy non-viable
* Twins or higher multiple pregnancies
* Outside age range
* Diabetes or pre-existing hypertension, chronic kidney disease or autoimmune disorders

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Healthy pregnant women scheduled for elective Caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
6-hydroxymelatonin sulphate in serum | 24 hours after delivery
  Change in serum 6-hydroxymelatonin sulphate levels after delivery

SECONDARY OUTCOMES:
6-hydroxymelatonin sulphate in serum | Immediately after delivery
  Serum 6-hydroxymelatonin sulphate levels in umbilical cord blood after delivery
6-hydroxymelatonin sulphate in placental tissue | Immediately after delivery
  Serum 6-hydroxymelatonin sulphate levels in placental tissue after delivery

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Aberdeen/NHS Grampian, Aberdeen, If Already Stated Select NOT Listed
  - Aberdeen Maternity Hospital, Ellon, Lowland Scotland

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests for access to anonymous IPD (biochemical data) will be considered